CLINICAL TRIAL: NCT00518401
Title: Phase I Study of A Combination Stem Cell Therapy is Safe and Feasible in the Development of Mature Stable Vessels in Ischemic Limbs
Brief Title: Combination Stem Cell Therapy for the Treatment of Severe Leg Ischemia
Acronym: mesendo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Gabriel P. Lasala, MD, TCA Cellular Therapy, LLC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-01-I
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-02

CONDITIONS: Critical Limb Ischemia; Peripheral Vascular Disease
Keywords: A hypoperfusion of the blood through a leg; Stem cells; Stem cell transplantation; Stem cell autologous transplantation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Mesendo — Intramuscular injection of 0.5 cc per site of the combination stem cell mixture in approximately 40 different ischemic sites of the gastrocnemius area of the calf.

SUMMARY:
The purpose of this research study is to determine if the transplant of a combination of stem cells obtained from the bone marrow of the same patient will contribute to the formation of new blood vessels in the severely diseased ischemic limb (leg). In this study the safe use of this combination of stem cells and its effects on making new blood vessels will be evaluated.

Limb Ischemia (LI) is a severe obstruction of the arteries which seriously decreases blood flow to the extremities (mainly feet and legs) and has progressed to the point of severe pain and even skin ulcers or sores.

LI needs comprehensive treatment since the condition will not improve on its own. The overall goal of treatment is to reduce the pain and increase blood flow to improve symptoms or save the leg or feet. In many cases, current options for treatment including medications, surgery or endovascular procedures have not been successful.

In the last few years, investigators have explored therapies aimed to increase blood flow to the ischemic vessels by transplanting cells that will promote the development of new vessels in the diseased leg.

The study hypothesis is based on the concept that the process of formation of new blood vessels is complex and requires the participation of several types of stem cells and growth factors. The lack of any of these components will produce vessels which are immature and unable to provide appropriate blood supply to the leg.

Patients eligible to participate in this study are those suffering from poor circulation or severe leg blockages, which are not candidates for surgical procedures.

Once the mixture of stem cells is prepared and the patient's bone marrow is ready, cells will be transplanted into the calf muscle of the diseased leg. Clinical studies to evaluate if the transplant works and is safe will be performed up to 1 year after cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Males or females older than 18 years of age.
* Limb ischemia with ABI of £ 0.6 in the index lower extremity in two consecutive examinations done at least 1 week apart.
* Limb ischemia with resting ischemic pain and/or non-healing ulcers.
* Patients not considered candidates for surgical or percutaneous revascularization, due to poor target vessels, inability to cross total occlusions, or a morbidity which precludes general anesthesia

Exclusion Criteria:

* Inability to provide informed consent.
* Previous angiogenic therapy.
* Known sensitivity to gentamycin and/or amphotericin B.
* Use or expected use of antineoplastic drugs.
* Any illness which might affect the patient's survival after enrollment in the protocol.
* Any illness or significant laboratory abnormality, which in the investigator's judgment will interfere with the patient's ability to comply with the protocol, compromise the patient's safety, or interfere with the interpretation of the study results.
* No evidence of acute infection - WBC > 15000.
* WBC < 4000.
* Serum Creatinine > 3.0 mg/dL.
* Pregnant women or women planning to become pregnant.
* Recent myocardial infarction within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel P. Lasala, MD, FACC, Principal Investigator — TCA Cellular Therapy
Locations (1):
- TCA Cellular Therapy, Covington, Louisiana, United States